CLINICAL TRIAL: NCT01980914
Title: Impact of Hypoglycemia on Cardiac Function in Elderly Patients With Diabetes
Brief Title: Hypoglycemia (Low Blood Sugar) and the Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Icentia UK (Industry)
Responsible Party: Principal Investigator, Graydon Meneilly, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H13-02734; unfunded (Other: UBC)
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Hypoglycemia; Type 2 Diabetes
Keywords: hypoglycemia; type 2 diabetes; insulin glargine; cardiac function; myocardial ischemia; cardiac rhythm; autonomic cardiovascular function
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 2; Myocardial Ischemia

STUDY DESIGN:
Intervention Model Description: We propose a pilot study in 20 patients over age 70 who have had type 2 diabetes for at least 5 years and are being treated with insulin All patients will have a BMI of between 20 and 35 Kg/M2, and an A1C between 7 and 8.5 %. All patients will have well controlled hypertension and hyperlipidemia. Patients with a GFR less than 40ml/min, poorly controlled CHF and active coronary artery disease or cerebrovascular disease will be excluded, although a past history of CAD or stroke will not result in exclusion
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 2 diabetes group (Experimental): Patients over age 70 who have had type 2 diabetes for at least 5 years and are being treated with insulin. All patients will have a BMI of between 20 and 35 Kg/M2, and an A1C between 7 and 8.5 %.
  Interventions: Device: iPro2 glucose sensor attachment

INTERVENTIONS:
Device: iPro2 glucose sensor attachment — At the same time the glucose sensor is started, a trained research nurse will connect the patient to an Icentia CardioSTAT, a continuous ambulatory ECG cardiac monitor.
  Other Names: Icentia CardioSTAT

SUMMARY:
The risk of hypoglycemia (low blood sugar) associated with the treatment of diabetes increases with age. Hypoglycemia is a common reason for admission to hospital for older patients with diabetes. Older patients are often unaware that their blood sugar is low and asymptomatic hypoglycemia, as assessed by continuous blood sugar monitoring, is frequent in the elderly. There is also evidence that older people with diabetes are more likely to develop cardiovascular events such a heart attack and more likely to die suddenly when compared to older people without diabetes. It is possible that low blood sugar levels contribute to the increased frequency of these events, but this possibility has never been studied. The purpose of this study is to assess how frequently low blood sugar occurs in older patients with diabetes and to see if low blood sugars adversely affect heart function in these patients.

DETAILED DESCRIPTION:
Investigators propose a pilot study in 20 patients over age 70 who have type 2 diabetes and are being treated with insulin. These patients will be enrolled from the elderly diabetes clinic at Vancouver General Hospital. Patients will be asked to come to the Gerontology research laboratory in the Research Pavilion at Vancouver General Hospital. A trained research nurse will instrument each patient with an iPro2 glucose sensor (Medtronic Canada). These sensors reliably and continuously measure blood glucose for periods of up to 7 days. Briefly, the skin will be swabbed with a disinfectant and a small catheter will be inserted subcutaneously. This needle will be attached to a glucose sensor. Patients will wear this sensor for 6 days. Patients will measure their glucose using a glucometer 4 times each day during this period and will also be given a log book to keep track of glucose values. Patients will also be asked to record any symptoms of hypoglycemia. At the end of 6 days the sensor will be removed.

At the same time the glucose sensor is started, a trained research nurse will connect the patient to a single use CardioSTAT ECG recorder. The archived ECG waveforms will be downloaded for QT and T-wave alternans analysis. The heart rate and QT interval will be measured at baseline and the end of each interval from the digitized ECG.

Patients and relevant family will be provided with in person education regarding the function and use of the monitor, implications for bathing and sleep, and contact information for troubleshooting. Patients will be asked to change the leads at home twice during the 6 days of the study. Patients will be asked to keep a log book of any cardiac symptoms during the 6 days of the study, as well as their activities. The glucose and CardioSTAT monitor will undergo time synchronization to ensure ability to do correlative analysis.

This is a feasibility pilot to establish preliminary data for analysis. The CardioSTAT monitor will allow assessment of cardiac arrhythmias, myocardial ischemia and cardiovascular autonomic function. The results from the glucose sensor and the CardioSTAT monitor will be correlated and compared to each other to determine if hypoglycemia has an adverse effect on heart function. Hypoglycemia is likely to induce autonomic responses captured on the CardioSTAT monitor and concordant ischemic S-T segment changes if coronary disease is present. It may also detect any resultant arrhythmias, although ischemic arrhythmias are uncommon in 6 days of monitoring. If investigators determine that hypoglycemia has negative effects on cardiac function, investigators may able to design treatments that would prevent these effects from happening in the future.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old and over
* had type 2 diabetes for at least 5 years
* treated with insulin glargine.
* BMI of between 20 and 35 Kg/M2,
* A1c between 7 and 8.5 %.
* well controlled hypertension and hyperlipidemia.

Exclusion Criteria:

* cannot speak english or give informed consent, or cognitive impairment
* glomerular filtration rate (GFR) less than 40ml/min,
* poorly controlled Chronic Heart Failure
* active coronary artery disease
* active cerebrovascular disease although a past history of CAD or stroke will not results in exclusion.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graydon S Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health Research Institute (VCHRI/VCHA) site -Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Patients: Patients over age 70 who have had type 2 diabetes for at least 5 years and are being treated with insulin. All patients will have a BMI of between 20 and 35 Kg/M2, and an A1C between 7 and 8.5 %. All patients will have well controlled hypertension and hyperlipidemia
Period: Overall Study
Arm/Group | Diabetic Patients
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only 11 participants were enrolled and 1 withdrew due to skin irritation
Groups:
- Diabetic Patients: We are aim to recruit group of 20 diabetic patients with type 2 diabetes over age 70, who are being treated with insulin.
  However, only 11 patients were enrolled.
  1 subject had experienced AE due to to skin irritation. 11 subjects have completed study.
Arm/Group | Diabetic Patients
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: Only 11 participants were enrolled, 1 withdrew due to skin irritation.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.4 (1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only 11 participants were enrolled, 1 withdrew due to skin irritation.
  Participants
    Female | 4
    Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Only participants from Vancouver area were invited to participate.
  Participants
    Canada | 11
Subjects with type 2 diabetes over age 70 [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hypoglycemia (Blood Sugar Level <70 mg/dl
Description: Track hypoglycemia with continuous glucose monitor. Subjects had measured their glucose using a glucometer 4 times each day during this period and were also got a log book to keep track of glucose values. They were also asked to record any symptoms of hypoglycemia. At the end of 6 days the sensor was removed.
Time Frame: 6 days
Population: Only participants who completed the study were analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Diabetic Patients: We are aim to recruit group of 20 diabetic patients with type 2 diabetes over age 70, who are being treated with insulin.
  However, only 11 patients were enrolled.
  1 subject withdrew after 24 hours due to skin irritation. 10 subjects have completed study.
Arm/Group | Diabetic Patients
Number analyzed (Participants) | 11
Participants | 11

2. Secondary Outcome: Alteration in Cardiac Rhythm
Description: To determine if there is a correlation between hypoglycemia and cardiac rhythm, alterations in cardiovascular autonomic function and myocardial ischemia.
Time Frame: 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Group
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse event date were collected during study period of up to 7 days when glucose sensors were attached.
Arm/Group | Diabetic Patients
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic Patients (N=11)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) — Skin irritation after glucose sensor was attached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT01980914/Prot_SAP_000.pdf